CLINICAL TRIAL: NCT01184300
Title: ReAssessment of Anti-Platelet Therapy Using an InDividualized Strategy Based on GENetic Evaluation (The RAPID GENE Study)
Brief Title: ReAssessment of Anti-Platelet Therapy Using an InDividualized Strategy Based on GENetic Evaluation
Acronym: RAPID GENE
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Collaborators: Spartan Bioscience Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HC-9427-U0143-43C
Record Dates: First submitted 2010-08-17; First posted 2010-08-18 (Estimated); Last update posted 2011-11-11 (Estimated); Status verified 2011-11

CONDITIONS: Stable Coronary Artery Disease; Acute Coronary Syndrome; Percutaneous Coronary Intervention
Keywords: CYP2C19*2; Pharmacogenomics; Clopidogrel; Prasugrel; Percutaneous Coronary Intervention
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Prasugrel Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rapid Genotyping (Experimental): Patients randomized to the Rapid Genotyping arm will have their CYP2C19*2 carrier status determined at the time of percutaneous coronary intervention with subsequent alteration in anti-platelet therapy for *2 carriers.
  Interventions: Genetic: Point-of-care genetic screening with subsequent prasugrel administration to CYP2C19*2 carriers
- Standard Therapy (No Intervention): Patients randomized to the Standard Therapy arm will not undergo genotyping at the time of percutaneous coronary intervention. All patients will receive clopidogrel 75 mg daily for 1 week. At the end of the 1 week period, their CYP2C19*2 carrier status will be verified.

INTERVENTIONS:
Genetic: Point-of-care genetic screening with subsequent prasugrel administration to CYP2C19*2 carriers — Patients found to carry the CYP2C19*2 allele will receive prasugrel 10 mg daily for 1 week. Non-carriers will receive clopidogrel 75 mg daily.
  Other Names: Prasugrel (Effient)
  Arms: Rapid Genotyping

SUMMARY:
The objective of the RAPID GENE study is to evaluate the feasibility, efficacy and safety of a pharmacogenomic approach to anti-platelet therapy following coronary artery stenting using a CYP2C19*2 point-of-care genetic test.

DETAILED DESCRIPTION:
Effective medical treatment following acute coronary syndromes and percutaneous coronary intervention (PCI) consists of dual anti-platelet therapy with aspirin and clopidogrel. Despite this treatment approach, a substantial portion of patients continue to experience an increased rate of subsequent adverse cardiovascular events including death, myocardial infarction, and stent thrombosis. This persistent vulnerability has been associated with inadequate platelet inhibition in response to clopidogrel administration, a phenomenon referred to as clopidogrel resistance. Although multiple variables have been implicated in clopidogrel resistance, mounting evidence suggests a crucial role for the loss-of-function CYP2C19*2 genetic variant. Presence of the *2 allele has been associated with a 1.5- to 6-fold increased risk of cardiovascular death, myocardial infarction, and stent thrombosis following PCI in patients treated with clopidogrel. These findings, recently bolstered by a meta-analysis, led the American Food and Drug Administration to issue a boxed warning for clopidogrel stating that poor metabolizers may not receive the full benefit of the drug. Consequently, experts have begun to advocate for routine genotyping in the context of dual anti-platelet therapy following PCI. A personalized approach to dual anti-platelet therapy following PCI is feasible given the presence of treatment alternatives such as prasugrel that are capable of overcoming clopidogrel resistance. Selective administration of prasugrel to patients at increased risk of clopidogrel resistance has the potential to successfully minimize adverse ischemic events, while simultaneously minimizing associated bleeding events and health care costs. A prospective pharmacogenomic approach to anti-platelet therapy has been previously hampered by limited access and the time-delay associated with genetic testing. The development of a point-of-care CYP2C19*2 genetic test that requires minimal training to operate carries the potential to overcome these obstacles and may facilitate the incorporation of pharmacogenomic strategies into routine clinical practice.

Patients receiving percutaneous coronary intervention in the context of non-ST elevation acute coronary syndromes and stable coronary artery disease will be randomized to either a rapid genotyping strategy or standard therapy. Patients in the Rapid Genotyping arm will be screened for the presence of the CYP2C19*2 allele using a point-of-care genetic test. Carriers of the *2 allele will receive prasugrel 10 mg daily for 1 week. Non-*2 carriers in the Rapid Genotyping arm and all patients in the Standard Therapy arm will receive clopidogrel 75 mg daily. At the end of the 1 week period, efficacy of the treatment strategies will be evaluated using VerifyNow platelet function testing.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females between the ages of 18 and 75 years
* Patients undergoing percutaneous coronary intervention in the context of a non-ST-elevation acute coronary syndrome or stable coronary artery disease
* Able to provide informed consent
* Able to comply with assigned treatment strategy and attend 1 week follow-up visit

Exclusion Criteria:

* Receiving anti-platelet therapy other than aspirin and clopidogrel
* Receiving anti-coagulation with warfarin
* History of stroke or transient ischemic attack
* Platelet count < 100 000/μL
* Known Bleeding Diathesis
* Hematocrit <32% or >52%
* Severe Liver Dysfunction
* Renal Insufficiency (Creatinine Clearance < 30ml/min)
* Pregnant females

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2010-08; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Clopidogrel response status as measured by the VerifyNow P2Y12 assay (Accumetrics, San Diego, CA) in CYP2C19*2 carriers. | 1 week
  Response status defined in P2Y12 Reaction Units (PRU) and percent platelet inhibition.

SECONDARY OUTCOMES:
Concordance of point-of-care genetic screening with laboratory based genotyping methods | 1 week
Composite of death from cardiovascular causes, non-fatal myocardial infarction, and re-hospitalization | 1 week and 6 months
Bleeding risk | 1 week and 6 months
  Defined by TIMI major/minor
Incidence of stent thrombosis | 1 week and 6 months
  ARC definitions
Feasibility of point-of-care genotyping in randomized setting | 1 week
Influence of Alternate CYP2C19 variants on outcomes | 1 week and 6 months
  CYP2C19 - functional polymorphisms

CONTACTS AND LOCATIONS:
Overall Officials: Derek Y.F. So, MD, Principal Investigator — Ottawa Heart Institute Research Corporation; Jason D. Roberts, MD, Study Director — Ottawa Heart Institute Research Corporation
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada

REFERENCES:
- [Background] Damani SB, Topol EJ. The case for routine genotyping in dual-antiplatelet therapy. J Am Coll Cardiol. 2010 Jul 6;56(2):109-11. doi: 10.1016/j.jacc.2010.03.029. Epub 2010 May 13. PMID 20471193
- [Background] Hulot JS, Collet JP, Silvain J, Pena A, Bellemain-Appaix A, Barthelemy O, Cayla G, Beygui F, Montalescot G. Cardiovascular risk in clopidogrel-treated patients according to cytochrome P450 2C19*2 loss-of-function allele or proton pump inhibitor coadministration: a systematic meta-analysis. J Am Coll Cardiol. 2010 Jul 6;56(2):134-43. doi: 10.1016/j.jacc.2009.12.071. PMID 20620727
- [Background] Mega JL, Close SL, Wiviott SD, Shen L, Hockett RD, Brandt JT, Walker JR, Antman EM, Macias W, Braunwald E, Sabatine MS. Cytochrome p-450 polymorphisms and response to clopidogrel. N Engl J Med. 2009 Jan 22;360(4):354-62. doi: 10.1056/NEJMoa0809171. Epub 2008 Dec 22. PMID 19106084
- [Background] Mega JL, Close SL, Wiviott SD, Shen L, Hockett RD, Brandt JT, Walker JR, Antman EM, Macias WL, Braunwald E, Sabatine MS. Cytochrome P450 genetic polymorphisms and the response to prasugrel: relationship to pharmacokinetic, pharmacodynamic, and clinical outcomes. Circulation. 2009 May 19;119(19):2553-60. doi: 10.1161/CIRCULATIONAHA.109.851949. Epub 2009 May 4. PMID 19414633
- [Background] Price MJ, Endemann S, Gollapudi RR, Valencia R, Stinis CT, Levisay JP, Ernst A, Sawhney NS, Schatz RA, Teirstein PS. Prognostic significance of post-clopidogrel platelet reactivity assessed by a point-of-care assay on thrombotic events after drug-eluting stent implantation. Eur Heart J. 2008 Apr;29(8):992-1000. doi: 10.1093/eurheartj/ehn046. Epub 2008 Feb 10. PMID 18263931
- [Background] Trenk D, Hochholzer W, Fromm MF, Chialda LE, Pahl A, Valina CM, Stratz C, Schmiebusch P, Bestehorn HP, Buttner HJ, Neumann FJ. Cytochrome P450 2C19 681G>A polymorphism and high on-clopidogrel platelet reactivity associated with adverse 1-year clinical outcome of elective percutaneous coronary intervention with drug-eluting or bare-metal stents. J Am Coll Cardiol. 2008 May 20;51(20):1925-34. doi: 10.1016/j.jacc.2007.12.056. PMID 18482659
- [Background] Sibbing D, Stegherr J, Latz W, Koch W, Mehilli J, Dorrler K, Morath T, Schomig A, Kastrati A, von Beckerath N. Cytochrome P450 2C19 loss-of-function polymorphism and stent thrombosis following percutaneous coronary intervention. Eur Heart J. 2009 Apr;30(8):916-22. doi: 10.1093/eurheartj/ehp041. Epub 2009 Feb 4. PMID 19193675
- [Derived] Roberts JD, Wells GA, Le May MR, Labinaz M, Glover C, Froeschl M, Dick A, Marquis JF, O'Brien E, Goncalves S, Druce I, Stewart A, Gollob MH, So DY. Point-of-care genetic testing for personalisation of antiplatelet treatment (RAPID GENE): a prospective, randomised, proof-of-concept trial. Lancet. 2012 May 5;379(9827):1705-11. doi: 10.1016/S0140-6736(12)60161-5. Epub 2012 Mar 29. PMID 22464343